CLINICAL TRIAL: NCT02130830
Title: Topical Anesthesia Versus Placebo to Decrease Post Procedure Pain in Rubber Band Ligation for the Treatment of Grade I - III Symptomatic Internal Hemorrhoids. A Single Institution, Double Blinded, Placebo Controlled Trial.
Brief Title: Topical Anesthesia Versus Placebo to Decrease Pain in Rubber Band Ligation for Treatment of Internal Hemorrhoids
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: 14-038
Record Dates: First submitted 2014-05-01; First posted 2014-05-05 (Estimated); Last update posted 2016-08-02 (Estimated); Status verified 2016-08

CONDITIONS: Hemorrhoids; Pain
Keywords: hemorrhoids; Rubber band ligation; pain
MeSH Terms: conditions — Hemorrhoids; Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Topical anesthesia (Experimental): Application of topical 2,5% lidocaine + 2,5% prilocaine gel to the anal canal before the procedure
  Interventions: Drug: Topical 2,5% lidocaine + 2,5% prilocaine gel
- Placebo (Placebo Comparator): Application of placebo gel into the anal canal before the procedure
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Topical 2,5% lidocaine + 2,5% prilocaine gel — The topical gel is administered in the anal canal at the moment of the anoscopy
  Arms: Topical anesthesia
Drug: Placebo — Placebo gel to mimic topical anesthesia administered in the anal canal at the moment of the anoscopy
  Arms: Placebo

SUMMARY:
Rubber band ligation is a simple and effective procedure for the management of hemorrhoidal disease. However, 90% of patients have some degree of discomfort associated with the procedure and up to 40% develop clinically significant pain. Some studies have used local anesthesia to reduce pain with promising results, but the use of topical anesthesia has not been reported before.

The investigators hypothesize that the use of topical anesthesia before rubber band ligation significantly reduces post procedure pain.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic grade I - III hemorrhoidal disease

Exclusion Criteria:

* Chronic liver disease
* Use of class 3 antiarrythmics
* Coagulopathy
* Grade IV hemorrhoidal disease
* Inflammatory bowel disease
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2014-05; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Pain measured in analog visual scale | up to 72 hours post procedure

SECONDARY OUTCOMES:
Procedure morbidity | up to 30 days post procedure

OTHER OUTCOMES:
Pain measured in visual analog scale in subgroups | up to 72 hours

CONTACTS AND LOCATIONS:
Overall Officials: Gellona Jose, MD, Principal Investigator — Pontificia Universidad Catolica de Chile; Bellolio Felipe, MD, Study Chair — Pontificia Universidad Catolica de Chile
Locations (1):
- Hospital Clínico Universidad Católica de Chile, Santiago, Santiago Metropolitan, Chile